CLINICAL TRIAL: NCT03872024
Title: Performances Evaluation of New FibroScan Probes Dedicated to Morbidly Obese Patients - NEO Study
Brief Title: Performances Evaluation of New FibroScan Probes Dedicated to Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M137
Record Dates: First submitted 2019-02-19; First posted 2019-03-12 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Obesity, Morbid; Liver Fibrosis
MeSH Terms: conditions — Obesity, Morbid; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morbidly obese adult patients (Experimental): Only one group of patients in the study: morbidly obese adult patients who will have an examination with the XXL probe prototype of the FibroScan 630 Research Model
  Interventions: Device: For the first 60 patients: 3 XXL probe prototypes of the FibroScan 630 Research Model; Device: From patient 61 to patient 120: 1 XXL probe prototype of the FibroScan 630 Research Model

INTERVENTIONS:
Device: For the first 60 patients: 3 XXL probe prototypes of the FibroScan 630 Research Model — After the patient informed consent form signature and during the patient pre-operative routine hospitalization, the following examinations will be done:
  * An ultrasound examination
  * One examination with the FibroScan® 430 mini fitted with the XL+ probe (commercial reference)
  * Three examinations with the FibroScan® 630 Expert - Research model fitted with the 3 XXL probe prototypes.
Device: From patient 61 to patient 120: 1 XXL probe prototype of the FibroScan 630 Research Model — After the patient informed consent form signature and during the patient pre-operative routine hospitalization, the following examinations will be done:
  * An ultrasound examination
  * One examination with the FibroScan® 430 mini fitted with the XL+ probe (commercial reference)
  * One examination with the FibroScan® 630 Expert - Research model fitted with 1 adjusted XXL+ probe prototype (H+F prototype probe).

SUMMARY:
Non-Alcoholic Fatty Liver is a common clinical and histological condition associated with metabolic syndrome in patients with and without excess body weight. It represents the most common cause of liver disease in the western world and it is characterized by an excess accumulation of fatty vacuole within hepatocytes.

Patients with non-alcoholic fatty liver disease (NAFLD) can progress to non-alcoholic steatohepatitis (NASH), and then into cirrhosis and its complications.

The prevalence of hepatic steatosis goes from 16 to 31% in the general population, from 50 to 80% in the obese population and up to 96% in morbidly obese patients. As the majority of obese individuals have NAFLD, non-invasive and widely applicable screening tools for the assessment of liver fibrosis and steatosis are needed. The detection in early stages is the main predictive factor of the long-term outcome.

Liver biopsy has traditionally been the gold standard for the assessment of patients with NAFLD, although the well-known limitations. Among the non-invasive tools available in the market, the FibroScan® (Echosens™, Paris, France) has been shown to be a useful tool for diagnosing fibrosis and steatosis in patients with suspected NAFLD. The FibroScan® is an ultrasound-based vibration-controlled transient elastography (VCTE™) device dedicated to liver stiffness measurement (LSM) and the controlled attenuation parameter (CAP).

Several clinical studies have shown the benefit of measuring hepatic stiffness with the FibroScan® in overweight/moderately obese persons. The ability to identify significant fibrosis and cirrhosis has been demonstrated in normal and overweight patients affected with chronic hepatitis B and C, biliary diseases, alcohol related liver disease and NAFLD.

However, subcutaneous fat attenuates the transmission of shear waves into the liver and the ultrasonic signals used to measure their speed of propagation. When scanning morbidly obese patients (BMI≥35 kg/m²) with the XL+ probe, unreliable results occur mainly due to obesity. Therefore, the XL probe has been enabled to expand the applicability of the FibroScan® but, the realization of the XL+ examination is still very difficult in the case of morbidly obese patients. This is why to reduce this failure rate, Echosens has worked on developing the XXL probe specifically for measuring the LSM in morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years old
* Patient must be able to give written informed consent
* Patient affiliated to a social security system
* Patients participating in the standard bariatric surgery care program (bariatric surgery criteria defined with BMI ≥ 40 kg / m² or patients with BMI ≥ 35 kg / m² and at least 1 associated co-morbidity

Exclusion Criteria:

* Patient with presence of ascites
* Patients with exclusion criteria for bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Liver biopsy: fibrosis stage from F0 to F4 with Kleiner (NASH CRN) scoring system | 12 months
  A liver biopsy will be performed during the bariatric surgery and will be sent to a centralized pathologist that will quantify the fibrosis and classify it from F0 to F4. Where F0 indicates the absence of fibrosis and F4 indicates cirrhosis.

SECONDARY OUTCOMES:
Number of valid measurements per probe higher than 8 | 12 months
  In order to be considered as a reliable exam, at least 8 valid measurements should be taken by the XL probe and the XXL prototype probes. Invalid measurements can appear when the probe connected to the FibroScan can't take a measurement for different reasons (distance skin to capsule very big, not good positioning of the probe….).
Liver Stiffness Measurement (LSM) from 1.5 to 75 kPa assessed with the FibroScan | 12 months
  The FibroScan stiffness measurement relies on the propagation of elastic waves to assess the stiffness of the liver: the faster elastic waves propagates within the liver, the stiffer the organ is. The final LSM value is the median of individual LSM values using the valid measurements and is expressed in kilo Pascal (kPa). Values obtained for the LSM with every probe will be assessed.
Controlled Attenuation Parameter (CAP) from 100 to 400 dB/m, assessed with the FibroScan | 12 months
  The intensity of ultrasonic signals received by the probe, which decrease as a function of depth and according to the medium, is measured:the CAP is the ultrasonic attenuation rate and is expressed in decibel per meter (dB/m). Values obtained for the CAP with every probe will be assessed.
Liver biopsy: steatosis grade from S0 to S3 with Kleiner (NASH CRN) scoring system | 12 months
  Measure and classify the steatosis grade (fat in the liver) by analyzing the liver biopsy. Where S0 represents the minimal steatosis grade (<5% hépatocytes with fat) and S3 indicates a steatosis with >66% hépatocytes with fat.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital la Pitié Salpêtrière, Paris, France